CLINICAL TRIAL: NCT05761444
Title: A Phase 4, Multicenter, Randomized, Open-label, Active-controlled Study to Evaluate the Effectiveness and Safety of Early add-on of Ezetimibe With Atorvastatin in Very High-risk Patients
Brief Title: Effectiveness and Safety Study of Early add-on of Ezetimibe With Atorvastatin in Very High-risk Patients
Acronym: BETTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OG-KORATO-001
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-10

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Very high-risk patients' Atherosclerotic cardiovascular disease (ASCVD)
MeSH Terms: conditions — Atherosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eze/Ato: Ezetimibe/Atorvastatin (Experimental): Participants will receive ezetimibe/atorvastatin 10/40 mg QD from Visit 2 (Day 1) to Visit 3 (Week 6). If the LDL-C target is reached (LDL-C < 55 mg/dL) at Visit 3, maintain the dose to Visit 4 (Week 12). If the LDL-C target level is not reached at Visit 3, dose is increased to ezetimibe/atorvastatin 10/80 mg QD from Visit 3 to Visit 4.
  Interventions: Drug: Atozet 10/40 mg or 10/80 mg
- Ato: Atorvastatin (Active Comparator): Participants will receive atorvastatin 40 mg QD from Visit 2 (Day 1) to Visit 3 (Week 6). If the LDL-C target is reached (LDL-C < 55 mg/dL) at Visit 3, maintain the dose to Visit 4 (Week 12). If the LDL-C target is not reached at Visit 3, dose is increased to atorvastatin 80 mg QD from Visit 3 to Visit 4.
  Interventions: Drug: Lipitor 40 mg or 80 mg

INTERVENTIONS:
Drug: Atozet 10/40 mg or 10/80 mg — Atozet 10/40 mg or 10/80 mg Dosage Formulation: Tablet Dosing Instructions: oral. Take 1 tablet daily
  Arms: Eze/Ato: Ezetimibe/Atorvastatin
Drug: Lipitor 40 mg or 80 mg — Lipitor 40 mg or 80 mg Dosage Formulation: Tablet Dosing Instructions: oral. Take 1 tablet daily
  Arms: Ato: Atorvastatin

SUMMARY:
This study aims to confirm the effectiveness of ezetimibe add-on therapy on LDL-C levels compared to atorvastatin monotherapy, especially in very high-risk patients. We intend to lay the foundation for a standard treatment for these patients through ezetimibe add on lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥ 30 years old.
2. Patients with very high-risk*: clinical or unequivocal on imaging ASCVD. ASCVD includes previous ACS (MI or UA), stable angina, coronary revascularization (percutaneous coronary intervention (PCI), coronary artery bypass graft surgery (CABG), and other arterial revascularization procedures), stroke and transient ischaemic attack (TIA), and peripheral arterial disease (Mach F 2020).
3. Patients (a) who failed to achieve their target LDL-C goals with low and/or moderate intensity statin mono therapy for ≥ 4 weeks or (b) who are statin-naïve or have not been on a stable (unchanged) statin regimen for at least 4 weeks prior to enrollment

   * rosuvastatin < 10 mg, atorvastatin < 40 mg, and all dose of pitavastatin, simvastatin, lovastatin, pravastatin, and fluvastatin (Team G 2020).
4. Patients with LDL-C levels ≥ 70 mg/dL
5. Patients who are willing to maintain TLC throughout the study.
6. Patients who are willing to provide written informed consent prior to study enrollment.

Exclusion Criteria:

1. Patients with hypersensitivity to ezetimibe, atorvastatin or any of its inactive ingredients.
2. Patients with active liver disease or unexplained persistent elevations of hepatic transaminase levels. (aspartate transaminase (AST) or alanine transaminase (ALT) > 3 x upper limit of normal (ULN)).
3. Patients who have predisposing conditions with muscle disease (i.e., rhabdomyolysis or myopathy) or neuromuscular disease.
4. Patients with myasthenia gravis.
5. Female patients who are pregnant or have a potential to be pregnant and nursing.
6. Patients who are taking glecaprevir and pibrentasvir.
7. Patients with hereditary problems of galactose intolerance, lapp lactase deficiency, or of glucose-galactose malabsorption.
8. Patients with disease known to influence serum lipids or lipoproteins excluding dyslipidemia.
9. Patients with a history of cancer within 5 years.
10. Patients whose life expectancy is less than 6 months due to their medical conditions.
11. Patients with any condition or situation that might pose a risk to the participant or interfere with participation in the study.
12. Patients who have received any investigational medicine within 12 weeks of written informed consent or are going to receive during the clinical trial period.
13. Patients who are judged to be difficult to conduct clinical trials according to the judgment of the investigator.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: WonYoung Lee, Study Director — Organon
Locations (7):
- South Korea (7):
  - Eunpyeong St. Mary's Hospital, Seoul, Eunpyeong-gu
  - Inje University Ilsan-Paik Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Keimyung University Dongsan Medical Center, Daegu, Gyeongsangbuk-do
  - Ulsan University Hospital, Ulsan, Gyeongsangnam-do
  - Chonnam National University Hospital, Gwangju, Jeollanam-do
  - Kangbuk Samsung Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 4, open-label, active-controlled study was conducted in very high-risk dyslipidemia participants at 8 centers in South Korea between 26 July 2023 and 15 October 2024.
Pre-assignment Details: The study consisted of a screening period (1 week), an treatment period (12 weeks), and an end-of-study assessment (at Week 12). A total of 137 participants were randomized and enrolled in the study.
Groups:
- Ezetimibe/Atorvastatin: Participants received ezetimibe/atorvastatin 10/40 milligram (mg) tablet orally once a day (QD) from Day 1 to Week 6.
  If the low-density lipoprotein cholesterol (LDL-C) target was reached <55 mg/deciliter (dL) at Week 6, the dose was maintained up to Week 12. If the LDL-C target was not reached at Week 6, dose was increased to ezetimibe/atorvastatin 10/80 mg QD from Week 6 to Week 12.
- Atorvastatin: Participants received atorvastatin 40 mg tablet orally QD from Day 1 to Week 6.
  If the LDL-C target was reached <55 mg/dL at Week 6, the dose was maintained up to Week 12. If the LDL-C target was not reached at Week 6, dose was increased to atorvastatin 80 mg QD from Week 6 to Week 12.
Period: Overall Study
Arm/Group | Ezetimibe/Atorvastatin | Atorvastatin
Started | 67 | 70
Treated | 67 | 69
Completed | 59 | 65
Not Completed | 8 | 5
Not completed — Protocol Violation | 2 | 1
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety analysis set (SAS) included all randomized participants who received at least 1 dose of study treatment.
Groups:
- Ezetimibe/Atorvastatin: Participants received ezetimibe/atorvastatin 10/40 mg tablet orally QD from Day 1 to Week 6.
  If the LDL-C target was reached <55 mg/dL at Week 6, the dose was maintained up to Week 12. If the LDL-C target was not reached at Week 6, dose was increased to ezetimibe/atorvastatin 10/80 mg QD from Week 6 to Week 12.
- Total: Total of all reporting groups
Arm/Group | Ezetimibe/Atorvastatin | Atorvastatin | Total
Number analyzed (Participants) | 67 | 69 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (10.07) | 64.7 (10.66) | 64.9 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 55 | 52 | 107
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 67 | 69 | 136
Low-Density Lipoprotein Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 98.1 (23.81) | 107.8 (34.14) | 103.0 (29.79)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Low-Density Lipoprotein Cholesterol at Week 6
Description: Blood samples were collected to determine the LDL-C values. The percentage change from baseline was defined as 100 x (LDL-C value at 6 weeks - LDL-C value at baseline)/LDL-C value at baseline. Baseline was defined as the last non-missing measurement taken prior to reference start date.
Time Frame: Baseline (Day 1) and Week 6
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study treatment and had a baseline assessment of LDL-C and at least 1 valid post baseline measurement of LDL-C.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Ezetimibe/Atorvastatin | Atorvastatin
Number analyzed (Participants) | 65 | 67
percentage change | -48.97 (2.71) | -27.75 (2.47)
Statistical Analysis 1: Comparison: Ezetimibe/Atorvastatin vs Atorvastatin; Test type: Other; p < 0.0001, ANCOVA — The analysis of covariance (ANCOVA) model with treatment group (ezetimibe/atorvastatin, atorvastatin) and history of statin administration (yes, no) as fixed effects and baseline LDL-C as a covariate; Least Squares (LS) mean difference = -21.22, 95% CI 2-sided [-29.26 to -13.19]

2. Secondary Outcome: Percentage of Participants Who Achieved Low-Density Lipoprotein Cholesterol Goal of <55 mg/dL at Weeks 6 and 12
Description: Blood samples were collected to determine the LDL-C values. Participants with LDL-C <55 mg/dL were identified. Percentages are rounded off to the hundredth decimal place.
Time Frame: Weeks 6 and 12
Population: The FAS included all randomized participants who received at least 1 dose of study treatment and had a baseline assessment of LDL-C and at least 1 valid post baseline measurement of LDL-C. Only participants with data collected at specific timepoints are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Ezetimibe/Atorvastatin | Atorvastatin
Number analyzed (Participants) | 65 | 67
percentage of participants
  Week 6 | 46.2 | 9.0
  Week 12: number analyzed (Participants) | 60 | 65
  Week 12 | 55.0 | 15.4

3. Secondary Outcome: Percentage of Participants Who Achieved Low-Density Lipoprotein Cholesterol Goal of <70 mg/dL at Weeks 6 and 12
Description: Blood samples were collected to determine the LDL-C values. Participants with LDL-C <70 mg/dL were identified. Percentages are rounded off to the hundredth decimal place.
Time Frame: Weeks 6 and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ezetimibe/Atorvastatin | Atorvastatin
Number analyzed (Participants) | 65 | 67
percentage of participants
  Week 6 | 78.5 | 38.8
  Week 12: number analyzed (Participants) | 60 | 65
  Week 12 | 85.0 | 58.5

4. Secondary Outcome: Percentage Change From Baseline in Low-Density Lipoprotein Cholesterol at Week 12
Description: Blood samples were collected to determine the LDL-C values. The percentage change from baseline was defined as 100 x (LDL-C value at 12 weeks - LDL-C value at baseline)/LDL-C value at baseline. Baseline was defined as the last non-missing measurement taken prior to reference start date.
Time Frame: Baseline (Day 1) and Week 12
Population: The FAS included all randomized participants who received at least 1 dose of study treatment and had a baseline assessment of LDL-C and at least 1 valid post baseline measurement of LDL-C. Only participants with data collected at baseline and Week 12 are reported.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Ezetimibe/Atorvastatin | Atorvastatin
Number analyzed (Participants) | 60 | 65
percentage change | -50.37 (2.60) | -34.41 (2.32)
Statistical Analysis 1: Comparison: Ezetimibe/Atorvastatin vs Atorvastatin; Test type: Other; p < 0.0001, ANCOVA — The ANCOVA model with treatment group (ezetimibe/atorvastatin, atorvastatin) and history of statin administration (yes, no) as fixed effects and baseline LDL-C as a covariate; LS mean difference = -15.96, 95% CI 2-sided [-23.56 to -8.36]

5. Secondary Outcome: Percentage Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C), Non-High-Density Lipoprotein Cholesterol (Non-HDL-C), Triglycerides, and Total Cholesterol at Weeks 6 and 12
Description: Blood samples were collected to determine the HDL-C, non-HDL-C, triglycerides, and total cholesterol values. The percentage change from baseline for HDL-C was defined as 100 x (HDL-C value at 6 or 12 weeks - HDL-C value at baseline)/HDL-C value at baseline. The percentage change from baseline for non-HDL-C was defined as 100 x (non-HDL-C value at 6 or 12 weeks - non-HDL-C value at baseline)/non-HDL-C value at baseline. The percentage change from baseline for triglycerides was defined as 100 x (triglycerides value at 6 or 12 weeks - triglycerides value at baseline)/triglycerides value at baseline. The percentage change from baseline for total cholesterol was defined as 100 x (total cholesterol value at 6 or 12 weeks - total cholesterol value at baseline)/total cholesterol value at baseline. Baseline was defined as the last non-missing measurement taken prior to reference start date.
Time Frame: Baseline (Day 1) and Weeks 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Ezetimibe/Atorvastatin | Atorvastatin
Number analyzed (Participants) | 65 | 67
percentage change
  Week 6: HDL-C | -2.44 (17.837) | -0.18 (17.479)
  Week 12: HDL-C: number analyzed (Participants) | 60 | 65
  Week 12: HDL-C | -2.15 (18.964) | -1.47 (17.163)
  Week 6: non-HDL-C: number analyzed (Participants) | 65 | 65
  Week 6: non-HDL-C | -35.36 (18.378) | -24.36 (21.625)
  Week 12: non-HDL-C: number analyzed (Participants) | 60 | 63
  Week 12: non-HDL-C | -39.97 (15.558) | -29.48 (18.422)
  Week 6: Triglycerides | -9.67 (40.806) | -4.94 (59.649)
  Week 12: Triglycerides: number analyzed (Participants) | 60 | 65
  Week 12: Triglycerides | -16.67 (31.948) | -1.49 (65.605)
  Week 6: Total cholesterol: number analyzed (Participants) | 65 | 65
  Week 6: Total cholesterol | -26.28 (14.692) | -18.51 (15.754)
  Week 12: Total cholesterol: number analyzed (Participants) | 60 | 63
  Week 12: Total cholesterol | -29.57 (13.563) | -22.18 (13.722)

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) at Weeks 6 and 12
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant administered a medicinal product and which does not necessarily have a causal relationship with that product. An SAE was defined as any AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. A TEAE was defined as AEs that first occurred or worsened in severity on or after the first administration of the study treatment during the treatment period.
Time Frame: From the first dose administration of the study treatment (Day 1) up to Week 6; From the first dose administration of the study treatment (Day 1) up to Week 12
Population: The SAS included all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ezetimibe/Atorvastatin | Atorvastatin
Number analyzed (Participants) | 67 | 69
Participants
  Week 6: Any TEAE | 9 | 8
  Week 6: Any TESAE | 3 | 2
  Week 12: Any TEAE | 15 | 13
  Week 12: Any TESAE | 4 | 3

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Event Leading to the Premature Discontinuation of the Study
Description: An AE was defined as any untoward medical occurrence in a clinical study participant administered a medicinal product and which does not necessarily have a causal relationship with that product. An SAE was defined as any AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. A TEAE was defined as AEs that first occurred or worsened in severity on or after the first administration of the study treatment during the treatment period.
Time Frame: as for outcome 6
Population: The SAS included all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ezetimibe/Atorvastatin | Atorvastatin
Number analyzed (Participants) | 67 | 69
Participants
  Week 6 | 2 | 2
  Week 12 | 3 | 2

ADVERSE EVENTS:
Time Frame: TEAEs are reported from the first dose administration of the study treatment (Day 1) up to end of the study, 12 weeks.
Description: The SAS included all randomized participants who received at least 1 dose of study treatment.
Arm/Group | Ezetimibe/Atorvastatin | Atorvastatin
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/69
Serious Adverse Events (participants affected / at risk) | 4/67 | 3/69
Other Adverse Events (participants affected / at risk) | 12/67 | 11/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe/Atorvastatin (N=67) | Atorvastatin (N=69)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe/Atorvastatin (N=67) | Atorvastatin (N=69)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
AST/ALT ratio abnormal (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT05761444/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT05761444/SAP_001.pdf